CLINICAL TRIAL: NCT07271979
Title: Liposomal Bupivacaine Versus Ropivacaine for Preperitoneal Infiltration Analgesia in Upper Abdominal Laparotomy: A Randomized Double-Blind Controlled Trial
Brief Title: Liposomal Bupivacaine Versus Ropivacaine for Preperitoneal Infiltration Analgesia in Upper Abdominal Laparotomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Jinying Zhang, Principal Investigator, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KYLL-202507-101-2
Record Dates: First submitted 2025-11-15; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Liposomal Bupivacaine; Preperitoneal Infiltration; Analgesia
MeSH Terms: conditions — Agnosia | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liposomal bupivacaine (Experimental): Prior to abdominal closure, the subject received a preperitoneal administration of liposomal bupivacaine at the surgical incision site. The total injection dose did not exceed 266 mg. A volume of 1 ml of the drug solution was administered per 1.5 cm of wound length per side.
  Interventions: Drug: Liposomal bupivacaine
- ropivacaine (Active Comparator): Prior to abdominal closure, the subject received a preperitoneal administration of 0.3% ropivacaine at the surgical incision site. A volume of 1 ml of the drug solution was administered per 1.5 cm of wound length per side.
  Interventions: Drug: ropivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — Upon abdominal closure following upper gastrointestinal open surgery, liposomal bupivacaine is administered preperitoneally along the surgical incision and diluted with normal saline according to the incision length.
  Arms: Liposomal bupivacaine
Drug: ropivacaine — Prior to abdominal closure following upper gastrointestinal open surgery, ropivacaine is administered preperitoneally at the surgical incision site and diluted with normal saline to a concentration of 0.3%.
  Arms: ropivacaine

SUMMARY:
Upper abdominal open surgery is associated with significant trauma, and postoperative pain management poses considerable challenges. The inflammatory response triggered by peritoneal incision and the transmission of visceral pain via the vagus nerve are key components of "surgical stress" and pain. A potential intervention strategy involves the local administration of anesthetic agents to suppress peritoneal overreaction and block the cascade of pro-inflammatory cytokines in related nerves. Liposomal bupivacaine, as a long-acting local anesthetic, may provide more prolonged postoperative analgesia compared to ropivacaine. Therefore, this trial aims to prospectively compare the analgesic efficacy and anti-inflammatory effects of the two drugs when administered as pre-closure preperitoneal infiltration. Secondary endpoints include opioid consumption, complication rates, and postoperative recovery indicators, to comprehensively evaluate their clinical value.

DETAILED DESCRIPTION:
Patients undergoing upper gastrointestinal open surgery often experience moderate to severe postoperative pain, which not only hinders early recovery but also significantly impairs their quality of life. Ideal postoperative analgesia requires a balance between efficacy and safety, and preperitoneal local anesthetic administration serves as an effective strategy to achieve this goal. Compared to conventional local anesthetics, liposomal bupivacaine-as a novel sustained-release formulation-enables continuous drug release, extending the analgesic duration to 48-72 hours. This study aims to compare the postoperative analgesic effects of preperitoneal injection of liposomal bupivacaine versus ropivacaine in patients undergoing upper gastrointestinal open surgery.

This study employs a randomized controlled design. Participants will be stratified based on the type of surgical incision (midline or subcostal) and randomized into groups using a computer-generated random seed with permuted block randomization (variable block sizes of 2, 4, and 6). Prior to abdominal closure during surgery, the experimental group will receive liposomal bupivacaine injections into the preperitoneal space on both sides of the wound, while the control group will receive ropivacaine injections. Apart from this intervention, both groups will maintain identical protocols for anesthesia induction, maintenance, and postoperative systemic analgesia to accurately evaluate the relative efficacy of the two local analgesic agents.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 70 years.
2. Scheduled for elective upper gastrointestinal open surgery.
3. Surgical approach involving either a subcostal or midline incision.
4. Incision length between 15 and 30 cm.
5. American Society of Anesthesiologists (ASA) physical status classification of I to III.

Exclusion Criteria:

1. ASA Physical Status Class greater than III.
2. Pre-existing chronic pain with long-term opioid use (for >1 year).
3. Significant hepatic or renal impairment, or underweight status, defined as:

   Estimated glomerular filtration rate (eGFR) of <40 mL/min/1.73m²; Child-Pugh Class C; Body Mass Index (BMI) <18.5 kg/m².
4. Known allergy or hypersensitivity to the investigational drug or any of its excipients.
5. Pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
postoperative pain score（NRS） | Day 1
  The Numeric Rating Scale (NRS) is an 11-point scale ranging from 0 to 10, where 0 represents "no pain" and 10 represents the "worst pain imaginable." Based on this, scores of 1-3 indicate mild pain, 4-6 indicate moderate pain requiring intervention, and 7-10 indicate severe pain necessitating urgent treatment. In this study, the investigators primarily assessed the incidence of an NRS score ≥ 4 within 24 hours postoperatively and the worst pain experienced by patients during that period.

SECONDARY OUTCOMES:
Time to First Rescue Analgesia and Number of Effective Patient-Controlled Intravenous Analgesia (PCIA) | Day 3
  The PCIA protocol (sufentanil 2 μg/kg in 100 mL saline, no background infusion, 3 mL bolus, 30-min lockout) was used. We recorded the time to first PCIA activation and the cumulative number of effective boluses within the first 72 postoperative hours.
the use of flurbiprofen axetil | Day 3
  the amount of rescue analgesic drugs flurbiprofen axetil used
postoperative adverse events | The first 3 postoperative days
  the incidence of nausea, vomiting, and vertigo after surgery
The Richards-Campbell Sleep Questionnaire | day 3
  It uses a 0-100 mm visual analog scale, with higher scores indicating better sleep quality.
Quality of Recovery-15 (QOR-15) scale | The first 3 postoperative days
  The scores from all 15 questions are summed to yield a total score ranging from 0 to 150, with a higher total score indicating a better quality of recovery for the patient.
Overall Benefit of Analgesia Score | The first three postoperative days
  This score is a patient-reported outcome measure for comprehensively evaluating the effectiveness of postoperative analgesic regimens, using a 29-point scale from 0 (best) to 28 (worst).
Changes in postoperative pain | The first 3 postoperative days
  Changes in pain scores (NRS) within the first 3 days postoperatively, including scores at rest at 6, 12, 24, 48, and 72 hours, as well as the peak pain level during this 3-day period.
hospital length of stay | From date of hospital admission until the date of discharge,assessed up to 15 days.
  The time between hospital admission and discharge
C-reactive protein | On the preoperative day and postoperative day 1
  The inflammatory marker of participants will be test after surgery
White Blood Cell Count and Differential | Day 1
  By analyzing the WBC profile-including both total count and cell type distribution-the inflammatory condition of a patient can be evaluated.
Postoperative Complications | One month after surgery
  The probability of patients acquiring pulmonary complications after surgery.

REFERENCES:
- [Background] Othman AH, Ahmed DG, Abd El-Rahman AM, El Sherif FA, Mansour S, Aboeleuon E. Effect of Preperitoneal Versus Epidural Analgesia on Postoperative Inflammatory Response and Pain Following Radical Cystectomy: A Prospective, Randomized Trial. Clin J Pain. 2019 Apr;35(4):328-334. doi: 10.1097/AJP.0000000000000679. PMID 30829734
- [Background] Colibaseanu DT, Osagiede O, Merchea A, Ball CT, Bojaxhi E, Panchamia JK, Jacob AK, Kelley SR, Naessens JM, Larson DW. Randomized clinical trial of liposomal bupivacaine transverse abdominis plane block versus intrathecal analgesia in colorectal surgery. Br J Surg. 2019 May;106(6):692-699. doi: 10.1002/bjs.11141. Epub 2019 Mar 28. PMID 30919948
- [Background] Pedrazzani C, Park SY, Conti C, Turri G, Park JS, Kim HJ, Polati E, Guglielmi A, Choi GS. Analgesic efficacy of pre-emptive local wound infiltration plus laparoscopic-assisted transversus abdominis plane block versus wound infiltration in patients undergoing laparoscopic colorectal resection: results from a randomized, multicenter, single-blind, non-inferiority trial. Surg Endosc. 2021 Jul;35(7):3329-3338. doi: 10.1007/s00464-020-07771-6. Epub 2020 Jul 6. PMID 32632489
- [Background] Gasanova I, Alexander J, Ogunnaike B, Hamid C, Rogers D, Minhajuddin A, Joshi GP. Transversus Abdominis Plane Block Versus Surgical Site Infiltration for Pain Management After Open Total Abdominal Hysterectomy. Anesth Analg. 2015 Nov;121(5):1383-8. doi: 10.1213/ANE.0000000000000909. PMID 26252171
- [Background] Beaussier M, El'Ayoubi H, Schiffer E, Rollin M, Parc Y, Mazoit JX, Azizi L, Gervaz P, Rohr S, Biermann C, Lienhart A, Eledjam JJ. Continuous preperitoneal infusion of ropivacaine provides effective analgesia and accelerates recovery after colorectal surgery: a randomized, double-blind, placebo-controlled study. Anesthesiology. 2007 Sep;107(3):461-8. doi: 10.1097/01.anes.0000278903.91986.19. PMID 17721249
- [Background] Tawfik MM, Mohamed YM, Elbadrawi RE, Abdelkhalek M, Mogahed MM, Ezz HM. Transversus Abdominis Plane Block Versus Wound Infiltration for Analgesia After Cesarean Delivery: A Randomized Controlled Trial. Anesth Analg. 2017 Apr;124(4):1291-1297. doi: 10.1213/ANE.0000000000001724. PMID 27984230
- [Background] Teo ZHT, Tey BLJ, Foo CW, Wong WY, Low JK. Intraoperative Celiac Plexus Block With Preperitoneal Infusion Reduces Opioid Usage in Major Hepato-pancreato-biliary Surgery: A Pilot Study. Ann Surg. 2021 Jul 1;274(1):e97-e99. doi: 10.1097/SLA.0000000000004883. PMID 33856374
- [Background] Ozer A, Yilmazlar A, Ozturk E, Yilmazlar T. Preperitoneal catheter analgesia is an effective method for pain management after colorectal surgery: the results of 100 consecutive patients. Local Reg Anesth. 2014 Oct 9;7:53-7. doi: 10.2147/LRA.S71476. eCollection 2014. PMID 25336988
- [Background] Alexander JC, Sunna M, Goldenmerry Y, Mootz A, O'Connor C, Ringqvist J, Bunker M, Joshi GP, Gasanova I. Comparison of transversus abdominis plane blocks with liposomal bupivacaine versus ropivacaine in open total abdominal hysterectomy. Proc (Bayl Univ Med Cent). 2022 Jun 30;35(6):746-750. doi: 10.1080/08998280.2022.2090798. eCollection 2022. PMID 36304627
- [Background] Ben-Saghroune H, Abdessadek M, Achour S, Kfal Y, El Bouazzaoui A, Kanjaa N, Sbai H. Assessment of the Safety and Efficiency of a Preperitoneal Continuous Infusion Using Bupivacaine after Abdominal Laparotomy in Digestive Carcinology. Anesthesiol Res Pract. 2023 Oct 10;2023:8842393. doi: 10.1155/2023/8842393. eCollection 2023. PMID 37854305
- [Background] Rawal N. Current issues in postoperative pain management. Eur J Anaesthesiol. 2016 Mar;33(3):160-71. doi: 10.1097/EJA.0000000000000366. PMID 26509324
- [Background] Sammour T, Kahokehr A, Soop M, Hill AG. Peritoneal damage: the inflammatory response and clinical implications of the neuro-immuno-humoral axis. World J Surg. 2010 Apr;34(4):704-20. doi: 10.1007/s00268-009-0382-y. PMID 20049432
- [Background] Baeriswyl M, Zeiter F, Piubellini D, Kirkham KR, Albrecht E. The analgesic efficacy of transverse abdominis plane block versus epidural analgesia: A systematic review with meta-analysis. Medicine (Baltimore). 2018 Jun;97(26):e11261. doi: 10.1097/MD.0000000000011261. PMID 29952997
- [Background] Ozturk E, Yilmazlar A, Coskun F, Isik O, Yilmazlar T. The beneficial effects of preperitoneal catheter analgesia following colon and rectal resections: a prospective, randomized, double-blind, placebo-controlled study. Tech Coloproctol. 2011 Sep;15(3):331-6. doi: 10.1007/s10151-011-0720-6. Epub 2011 Jul 19. PMID 21769617
- [Background] Joshi GP, Machi A. Surgical site infiltration: A neuroanatomical approach. Best Pract Res Clin Anaesthesiol. 2019 Sep;33(3):317-324. doi: 10.1016/j.bpa.2019.07.017. Epub 2019 Jul 25. PMID 31785717
- [Background] Mungroop TH, Bond MJ, Lirk P, Busch OR, Hollmann MW, Veelo DP, Besselink MG. Preperitoneal or Subcutaneous Wound Catheters as Alternative for Epidural Analgesia in Abdominal Surgery: A Systematic Review and Meta-analysis. Ann Surg. 2019 Feb;269(2):252-260. doi: 10.1097/SLA.0000000000002817. PMID 29781846
- [Background] Perniola A, Fant F, Magnuson A, Axelsson K, Gupta A. Postoperative pain after abdominal hysterectomy: a randomized, double-blind, controlled trial comparing continuous infusion vs patient-controlled intraperitoneal injection of local anaesthetic. Br J Anaesth. 2014 Feb;112(2):328-36. doi: 10.1093/bja/aet345. Epub 2013 Oct 31. PMID 24185607
- [Background] Mungroop TH, Veelo DP, Busch OR, van Dieren S, van Gulik TM, Karsten TM, de Castro SM, Godfried MB, Thiel B, Hollmann MW, Lirk P, Besselink MG. Continuous wound infiltration versus epidural analgesia after hepato-pancreato-biliary surgery (POP-UP): a randomised controlled, open-label, non-inferiority trial. Lancet Gastroenterol Hepatol. 2016 Oct;1(2):105-113. doi: 10.1016/S2468-1253(16)30012-7. Epub 2016 Jul 7. PMID 28404067